CLINICAL TRIAL: NCT00085384
Title: A Phase I/II Study to Evaluate the Optimum Dose of Pegylated-Interferon (PEG INTRON) in Patients With Platinum Resistant Ovarian, Peritoneal or Fallopian Tube Cancer
Brief Title: PEG-Interferon Alfa-2b in Treating Patients With Platinum-Resistant Ovarian Epithelial, Peritoneal, or Fallopian Tube Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID02-115; P50CA083639 (NIH); P30CA016672 (NIH); MDA-ID-02115 (Other: UT MD Anderson Cancer Center); CDR0000368964 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG-interferon alfa-2b (Experimental): Patients receive PEG-interferon alfa-2b (PEG IFN-α) subcutaneously (SC) on days 1, 8, 15, and 22.
  Interventions: Biological: PEG-interferon alfa-2b
- Arm II (Experimental): Patients receive PEG IFN-α SC (at a higher dose than in arm I) on days 1, 8, 15, and 22.
  Interventions: Drug: PEG-interferon alfa-2b
- Arm III (Experimental): Patients receive PEG IFN-α SC (at a higher dose than in arm II) on days 1, 8, 15, and 22.
  Interventions: Biological: PEG-interferon alfa-2b

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — Starting dose 1.0 mg/kg/week given subcutaneously
  Other Names: PEG-Intron
  Arms: PEG-interferon alfa-2b
Drug: PEG-interferon alfa-2b — Biological/Vaccine: PEG-interferon alfa-2b
  Dose 1.25 mg/kg/week given subcutaneously
  Other Names: PEG-Intron
  Arms: Arm II
Biological: PEG-interferon alfa-2b — Biological/Vaccine: PEG-interferon alfa-2b
  Dose 1.5 mg/kg/week given subcutaneously
  EG-Intron
  Other Names: PEG-Intron
  Arms: Arm III

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may interfere with the growth of cancer cells.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of PEG-interferon alfa-2b and to see how well it works in treating patients with ovarian epithelial, peritoneal, or fallopian tube cancer that is resistant to platinum-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimum biologic dose of PEG-interferon alfa-2b in patients with platinum-resistant ovarian epithelial, peritoneal, or fallopian tube cancer.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 3 different treatment arms.

* Arm I: Patients receive PEG-interferon alfa-2b (PEG IFN-α) subcutaneously (SC) on days 1, 8, 15, and 22.
* Arm II: Patients receive PEG IFN-α SC (at a higher dose than in arm I) on days 1, 8, 15, and 22.
* Arm III: Patients receive PEG IFN-α SC (at a higher dose than in arm II) on days 1, 8, 15, and 22.

In all arms, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for at least 28 days after study treatment.

PROJECTED ACCRUAL: A maximum of 75 patients will be accrued for this study within 19 months.

ELIGIBILITY:
Inclusion Criteria:

1. Women with platinum-resistant epithelial ovarian, fallopian tube or peritoneal cancer whose tumor test positive for IL-8 (>31.0 pg/ml), bFGF >7.0 pg/ml), or VEGF (>700 pg/ml). Resistance is defined as:

   1. Progression of disease during platinum chemotherapy, or
   2. Progression of disease within 6 months of completing platinum chemotherapy
   3. Failure to achieve a complete response, with persistent macroscopic disease, after 6 cycles of chemotherapy, if the last two cycles had no measurable change in disease status
2. Patients with a known hypersensitivity to platinum compounds who have failed a desensitization regimen, or who are not good candidates for desensitization are eligible.
3. Patients are limited to 4 prior chemotherapy regimens (all platinum and taxane regimens to be counted as one).
4. Patients must have measurable disease.
5. Women of any racial and ethnic group.
6. Zubrod performance status < 2.
7. Expected survival of > 12 weeks.
8. Patients must have adequate hepatic, renal, and bone marrow function, defined as serum creatinine < 2 mg/dl (estimated creatinine clearance 50 ml/min); total bilirubin < 2.0 X the upper limit of normal (ULN); alanine aminotransferase (ALT) < 2X ULN; fasting triglycerides < 800 mg/dL; white blood count (WBC) > 3,000/mm3 ; absolute neutrophil count (ANC) > 1,500/mm3; platelets > 100,000/mm3, hemoglobin > 9 g/dl.
9. At least three weeks must have elapsed from completion of chemotherapy.
10. Patient agrees not to use complementary alternative medications (e.g., shark cartilage).
11. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with the policies of the hospital. The only approved consent is appended to this protocol.

Exclusion Criteria:

1. Patients with borderline, low grade or low malignant potential tumors are not eligible.
2. Patients who are pregnant or lactating.
3. Concurrent chemotherapy, radiation therapy or surgery.
4. Concurrent, uncontrolled, medical or psychiatric disorders.
5. Patients with a known hypersensitivity to interferon.
6. Patients with severe cardiovascular disease (i.e. arrhythmias requiring chronic treatment or congestive heart failure) (NYHA classification III or IV).
7. Patients who have had interferon within the last 6 months.
8. Patients with overt psychosis or mental disability or otherwise incompetent to give informed consent.
9. Patients with a known autoimmune disorder.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-07; Primary Completion 2005-11 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Optimal Biologic Dose at 8 weeks | 8 weeks
  Optimum biologic dose of PEG Intron in patients with platinum-resistant ovarian, fallopian tube or peritoneal cancer whose tumors test positive for IL-8, BFGF, or VEGF.
Tumor Response | Every 2 -3 cycles (8 - 12 weeks)
  Each patient tumor response scored as either complete/partial response (CR/PR), stable disease (SD), or failure (F) at 8 weeks after initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Judith K. Wolf, MD, Study Chair — M.D. Anderson Cancer Center; Pedro T. Ramirez, MD, Study Chair — M.D. Anderson Cancer Center; Diane C. Bodurka, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org